CLINICAL TRIAL: NCT07134283
Title: The Effect of Preoperatively Initiated Cold Application on Postoperative Bleeding, Pain, and Functional Status in Total Knee Arthroplasty
Brief Title: Effect of Preoperative Cold Therapy on Early Postoperative Outcomes in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Omer Faruk Naldoven, Orthopedic Surgeon, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TABED 1-24-331
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Cryotherapy; Postoperative Pain Management; Opioid Consumption, Postoperative
Keywords: Total Knee Arthroplasty; Preoperative Cold Therapy; Cryotherapy; Postoperative Pain; Opioid Consumption; Knee Surgery; Drainage Output
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 into two parallel groups to receive either preoperative and postoperative cold therapy or only postoperative cold therapy.
Who Masked: Care Provider
Masking Description: Care providers such as nurses and physiotherapists responsible for postoperative rehabilitation and routine care were blinded to group allocation. Patients and outcome assessors were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative and Postoperative Cold Therapy (Experimental): Patients in this group received conventional cold therapy (gel pack at -17°C) both before and after surgery. Three sessions were applied preoperatively (20 minutes with 40-minute intervals), and postoperative therapy was performed identically to the control group (20 minutes on / 40 minutes off for 24 hours).
  Interventions: Procedure: Preoperative and Postoperative Cold Therapy with Gel Cold Pack
- Postoperative Cold Therapy Only (Active Comparator): Patients in this group received conventional cold therapy (gel pack at -17°C) after surgery only. Cold packs were applied to the knee region for 20 minutes with 40-minute intervals over a 24-hour postoperative period.
  Interventions: Procedure: Postoperative Cold Therapy with Gel Cold Pack

INTERVENTIONS:
Procedure: Preoperative and Postoperative Cold Therapy with Gel Cold Pack — Cold therapy was applied using a conventional gel cold pack , pre-cooled at -17°C for at least 2 hours. In the intervention group, cold application was performed three times before surgery (20 minutes per session with 40-minute intervals), and continued postoperatively for 24 hours with the same frequency. This protocol aimed to reduce pain, swelling, bleeding, and improve functional outcomes after total knee arthroplasty.
  Other Names: Traditional CryotherapY; Cold Application; Conventional Gel Pack
  Arms: Preoperative and Postoperative Cold Therapy
Procedure: Postoperative Cold Therapy with Gel Cold Pack — Cold therapy applied only in the postoperative period, for 24 hours, using the same method as the intervention group (20-minute applications with 40-minute breaks.
  Other Names: Traditional Cryotherapy; Cold Application; Conventional Gel Pack
  Arms: Postoperative Cold Therapy Only

SUMMARY:
This prospective, single-center, randomized controlled trial investigates the effects of preoperative cold therapy on early postoperative outcomes in patients undergoing unilateral primary total knee arthroplasty (TKA). A total of 208 patients were randomized into two groups: one receiving conventional cold therapy preoperatively and postoperatively, and the other receiving only routine postoperative cold therapy. Primary outcomes included postoperative pain (VAS), edema (thigh circumference), hemoglobin levels, drainage volume, opioid usage, Knee Society Scores (KSS), and presence of ecchymosis. The study demonstrated that initiating cold therapy before surgery significantly reduced postoperative drainage and opioid requirement, and delayed early edema progression. These findings suggest that the timing of cold therapy may influence recovery, highlighting a potentially beneficial approach to perioperative care in TKA.

DETAILED DESCRIPTION:
This prospective, single-center, randomized controlled study aims to evaluate the early postoperative effects of initiating cold therapy in the preoperative period in patients undergoing total knee arthroplasty (TKA). While cold therapy is routinely applied in the postoperative period to reduce pain, swelling, and inflammation, limited evidence exists regarding the impact of starting cold therapy before surgery. In this study, a total of 208 patients diagnosed with advanced degenerative knee osteoarthritis and scheduled for unilateral primary cemented TKA were randomly assigned to two groups: one receiving conventional gel-based cold therapy both preoperatively and postoperatively (intervention group), and one receiving only standard postoperative cold therapy (control group).

Cold therapy was applied using gel packs at -17°C for 20 minutes with 40-minute intervals. The intervention group received three preoperative sessions prior to surgery and continued postoperatively for 48 hours. The control group received only the postoperative protocol.

The primary outcomes were postoperative pain (measured using Visual Analog Scale - VAS), edema (thigh circumference), hemoglobin levels, drainage output at 24 hours, and opioid consumption during the first 48 hours. Secondary outcomes included Knee Society Scores (KSS), hospital stay duration, and presence of ecchymosis.

The results demonstrated that preoperative initiation of cold therapy significantly reduced postoperative drainage volume and opioid consumption, and showed a trend toward slower edema progression and lower pain scores in the early postoperative period. This study proposes a novel approach in perioperative management by emphasizing the importance of cold therapy timing, and provides evidence that beginning therapy preoperatively may enhance recovery outcomes after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* Diagnosed with advanced stage primary osteoarthritis of the knee
* Scheduled for unilateral primary total knee arthroplasty
* Provided written informed consent

Exclusion Criteria:

* Secondary osteoarthritis (e.g., post-traumatic, inflammatory arthritis)
* History of prior surgery on the affected knee
* Known hypersensitivity or intolerance to cold
* Comorbidities contraindicating cold therapy (e.g., diabetes mellitus, cold urticaria, peripheral vascular disease)
* Bleeding diathesis or on anticoagulant therapy
* History of severe hypertension or cardiovascular disease
* Active neurological or psychiatric disorder
* Allergy to medications used in the study protocol
* Refusal to participate in the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Scores for Pain | Preoperative, 8 Hours Postoperative, 24 Hours Postoperative, 48 Hours Postoperative
  Pain intensity was assessed using the Visual Analog Scale (VAS) at rest at four time points: Preoperative, 8 Hours Postoperative, 24 Hours Postoperative, 48 Hours Postoperative
  Scale Range: 0 (no pain) - 10 (worst imaginable pain)
  Directionality: Higher scores indicate worse pain
Postoperative Drainage Volume | First 24 hours after surgery
  Total amount of fluid collected in the Hemovac drainage system during the first 24 hours after total knee arthroplasty (TKA). This measure is used as an indicator of postoperative bleeding and local inflammation, comparing the effect of preoperative cold therapy.
Total Opioid Consumption in the First 48 Hours | First 48 hours after surgery
  Total opioid usage calculated as oral morphine equivalent in the first 48 hours after TKA. This includes all administered analgesics converted into oral morphine equivalent doses to evaluate pain control efficacy between study groups.
Hemoglobin Level Change | Preoperative, 8 Hours Postoperative, 24 Hours Postoperative, 48 Hours Postoperative
  Hemoglobin levels were recorded at four time points to evaluate perioperative blood loss: Preoperative, 8 Hours Postoperative, 24 Hours Postoperative, 48 Hours Postoperative
Knee Society Score (KSS) | Preoperative and 48 Hours Postoperative
  Functional outcomes were measured using the KSS scale, which includes pain, range of motion, and stability. Scores were compared preoperatively and at 48 hours postoperatively.
  Each component is scored from 0 to 100, with higher scores indicating better outcomes.
Thigh Circumference Measurement | Preoperative, 24 Hours Postoperative, 48 Hours Postoperative
  Thigh circumference was measured 1 cm proximal to the superior patella border with the knee in full extension, to assess postoperative swelling. Measurements were taken preoperatively, 24 hours postoperatively, and 48 hours postoperatively.

SECONDARY OUTCOMES:
Presence of Ecchymosis | 24 Hours Postoperative and 48 Hours Postoperative
  Ecchymosis was visually evaluated and recorded at 24 hours postoperatively and 48 hours postoperatively in both groups.
Need for Blood Transfusion | From Surgery Until Hospital Discharge(2 to 7 Days Postoperative)
  The number of patients who required postoperative blood transfusion was recorded and compared between the groups. The transfusion threshold was hemoglobin <8 g/dL in hemodynamically stable patients. The outcome will be assessed throughout the hospitalization period after surgery.
Length of Hospital Stay | Through Hospital Discharge (Estimated 2 to 7 Days Postoperative)
  The duration of hospitalization in days was recorded for each patient, from the day of surgery until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pieri L, Leggieri F, Bartoli D, Ponti M, Caparrini C, Baldini A. Preoperative knee joint hypothermia reduces inflammation and recovery time and increases range of motion after total knee arthroplasty: A randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2025 Dec;33(12):4312-4323. doi: 10.1002/ksa.12756. Epub 2025 Jul 2. PMID 40601965
- [Background] Chareancholvanich K, Keesukpunt W, Pornrattanamaneewong C, Narkbunnam R, Jarusriwanna A. Comparison of three cryotherapy techniques for early post-TKA pain control in terms of efficacy and patient satisfaction: a randomized controlled trial. Arthroplasty. 2025 Jan 8;7(1):5. doi: 10.1186/s42836-024-00287-7. PMID 39773549
- [Background] Thienpont E. Does advanced cryotherapy reduce pain and narcotic consumption after knee arthroplasty? Clin Orthop Relat Res. 2014 Nov;472(11):3417-23. doi: 10.1007/s11999-014-3810-8. Epub 2014 Jul 25. PMID 25059851
- [Background] Hawker G, Wright J, Coyte P, Paul J, Dittus R, Croxford R, Katz B, Bombardier C, Heck D, Freund D. Health-related quality of life after knee replacement. J Bone Joint Surg Am. 1998 Feb;80(2):163-73. doi: 10.2106/00004623-199802000-00003. PMID 9486722